CLINICAL TRIAL: NCT03344679
Title: A Comparative Study of Ultrasound Guided PECS Block Using Bupivacaine Adenosine Versus Bupivacaine Magnesium Sulphate: A Randomised Controlled Trial.
Brief Title: Adenosine and Magnesium Sulphate as Adjuvants for PECS Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MenoufiaU2015
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Breast Surgery
Keywords: Pectoral nerve block; Adenosine; Magnesium sulphate
MeSH Terms: interventions — Control Groups; Adenosine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Bupivacaine 0.25% for pectoral nerve block.
  Interventions: Drug: Bupivacaine 0.25%
- Adenosine (Other): Bupivacaine 0.25% with added Adenosine 12mg for pectoral nerve block.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Adenosine 12mg
- Magnesium sulphate (Other): Bupivacaine 0.25% with Magnesium sulphate 500 mg for pectoral nerve block.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Magnesium Sulphate 500 mg

INTERVENTIONS:
Drug: Bupivacaine 0.25% — Bupivacaine 0.25% for PECS block
  Other Names: Control group
Drug: Adenosine 12mg — Adenosine 12 mg for PECS block
  Other Names: Adenosine
  Arms: Adenosine
Drug: Magnesium Sulphate 500 mg — Magnesium sulphate 500 mg for PECS block
  Other Names: Magnesium sulphate
  Arms: Magnesium sulphate

SUMMARY:
Pectoral nerve block (PECS) has been used for post-operative pain relief in patients undergoing breast surgery. It has been shown that adenosine has an effect on pain modulation. Magnesium sulphate has been used as an adjuvant to local anaesthetics in many nerve block techniques. We hypothesised that adenosine may affect the PECS block quality. We aimed to compare the effect of adding adenosine to the local anaesthetic and compare its effect to magnesium sulphate when used for PECS block.

DETAILED DESCRIPTION:
The present study was conducted on 90 adult patients aged between 20 and 65 years old. Patients scheduled for modified radical mastectomy with axillary clearance surgery American Society of Anaesthetist (ASA) classes I, II, and III patients were included in the study.

Patients were randomly allocated into on of three groups according to the adjuvant used with the local anaesthetic, 30 patients in each group using a computerised program. All patients received PECS block. Group (C) received PECS block with 0.25% bupivacaine (control group), group (A) bupivacaine with added adenosine, and group (M) bupivacaine with added magnesium sulphate.

The local anaesthetic syringes were prepared by an independent anaesthetist. The researchers and the patients were blinded to the local anaesthetic adjuvant in the syringes. All patients received 30 ml local anaesthetic for PECS. The 30 ml local anaesthetic used for each patient contained bupivacaine hydrochloride 0.25%, bupivacaine hydrochloride 0.25% and 12 mg adenosine, and bupivacaine hydrochloride 0.25% and 500 mg magnesium sulphate for groups C, A, and M respectively.

Patients' demographic data were collected including age, BMI, ASA, and duration of surgery. In the post- anesthetic care unit (PACU) the visual analogue score (VAS) was assessed on arrival and then every 15 minutes. The duration and the quality of the block was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for modified radical mastectomy with axillary clearance surgery ASA classes I, II, and III patients were included in the study

Exclusion Criteria:

* 1) contraindications for regional anesthesia such as coagulopathy, local infection and fungating breast cancer, 2) history of allergy to the medications used in the study, 3) patient with history of drug abuse, 4) previous breast surgery except for diagnostic biopsies, 5) history of treatment for a chronic pain condition, 6) psychiatric disorder.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-22 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | First 24 hours after surgery
  Visual analogue scale is a scale from 1 to 10 where 1 is no pain and 10 is the worst pain the patient experienced.

SECONDARY OUTCOMES:
Analgesic requirement | First 24 hours after surgery
  The total amount of morphine (mg) consumed by patients.
PECS block duration. | First 24 hours after surgery
  The time from performing the block until the patient started to feel pain and the effect of the block faded.
Mean arterial blood pressure (mmHg) | Intra-operative (from induction of anaesthesia until the patient is awake)
  Mean arterial blood pressure reading.
Heart rate (beat/minute) | Intra-operative(from induction of anaesthesia until the patient is awake)
  The number of hear beats per minute

IPD SHARING:
Plan to Share IPD: No